CLINICAL TRIAL: NCT05517343
Title: Impact of Real-time Notification of Colonoscopic Optical Diagnosis on Patients' Anxiety and Depression After Polypectomy: a Randomized Control Trial
Brief Title: Impact of Real-time Notification of Colonoscopic Optical Diagnosis on Patients' Anxiety and Depression After Polypectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Chen-Ya Kuo, Attending physician, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJUH111207
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Neoplasms; Colonic Polyp; Anxiety; Depression; Colonoscopy
Keywords: colonoscopy; polypectomy; image enhanced endoscopy; endoscopic optical diagnosis
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label, prospective and parallel randomized controlled trial. This study planning to recruit outpatients from the age of 40 to 79 who are scheduled to undergo sedated colonoscopy and received polypectomy during the procedure. Participants will be randomized into "ordinary care group (explained at next scheduled clinic)" and "real-time notification group (explained immediately after colonoscopy)" in 1:1 ratio. Randomization will be based on a computer-generalized randomization list and stratified by gender and baseline anxiety degree of the participants. The level of anxiety, depression of the two groups will be measured by using the Taiwan version questionnaire of Hospital Anxiety and Depression Scale right before the next scheduled clinic for histological results and compared the difference between the two groups.
Masking Description: The participants, care providers, investigators and outcome assessors are not blinded to the assigned study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ordinary care (OC) (No Intervention): The participants of this arm received the endoscopic optical diagnosis, histological diagnosis of the resected colon polyps and the recommended surveillance colonoscopy schedule at next scheduled clinic visit (around 1 to 2 weeks later).
- Real-time notification (RTN) (Experimental): The participants of this arm received the endoscopic optical diagnosis of the resected colon polyps and the recommended surveillance colonoscopy schedule right after the sedated colonoscopy. Histological diagnosis will be informed at next scheduled clinic visit (around 1 to 2 weeks later).
  Interventions: Other: Real-time endoscopic optical diagnosis

INTERVENTIONS:
Other: Real-time endoscopic optical diagnosis — The participants assigned to real-time notification group will received the endoscopic diagnosis of the resected colorectal polyps and recommended surveillance colonoscopy schedule right after the sedated colonoscopy.
  Arms: Real-time notification (RTN)

SUMMARY:
The accuracy of endoscopic optical diagnosis for colorectal polyps has been approaching histological diagnosis after implementation of image enhancement endoscopic technologies. The real-time notification of possible nature of resected polyp after colonoscopy is expected to reduce the anxiety and depression level of the patients before the availability of histological diagnosis and improve their quality of life. We designed and conducted a randomized control trial to confirm this hypothesis.

DETAILED DESCRIPTION:
This is a single center, open-label, prospective and parallel randomized controlled trial. This study planning to recruit outpatients from the age of 40 to 79 who are scheduled to undergo sedated colonoscopy. Once eligible subjects were diagnosed of colorectal polyps during colonoscopy and received polypectomy, they will be randomized into "ordinary care group (explained at next scheduled clinic)" and "real-time notification group (explained immediately after colonoscopy)". The level of anxiety, depression of the two groups will be measured by using the Taiwan version questionnaire of Hospital Anxiety and Depression Scale (HADS) right before the next scheduled clinic for histological results and compared the difference between the two groups.This study is expected to determine the impact of real-time notification of colonoscopic optical diagnosis on patients' anxiety and depression after polypectomy, and provide evidence to improve post-polypectomy care.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥ 40 years and < 80 years
* Outpatients who prepare receiving sedated colonoscopy
* Subjects who have signed informed consent form of this study
* Informed consensus has been obtained that endoscopic resection should be performed if a colorectal polyp is found
* Eastern Cooperative Oncology Group (ECOG) performance status scale among 0 to 2

Exclusion Criteria:

* Subjects with any of the following prior history or current conditions:
* (a) Contraindications to colonoscopy
* (b) Major mental illnesses, e.g. major depressive disorder, schizophrenia, generalized anxiety disorder ...
* (c) Inflammatory bowel disease
* (d) Hereditary or non-hereditary polyposis syndrome, hereditary non-polyposis colorectal cancer
* (e) Uncured colorectal cancer
* (f) Active gastrointestinal bleeding
* (g) Pregnancy
* Subjects who do not received polypectomy during colonoscopy.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of definite anxiety cases | This outcome will be assessed right before the next scheduled clinic for histological results (around 1 to 2 weeks after polypectomy)..
  The level of anxiety of the two study arms will be measured by using the Taiwan version questionnaire of Hospital Anxiety and Depression Scale (HADS) right before the next scheduled clinic for histological results. The anxiety score of this questionnaire ranging from 0 to 21. Scored 0 to 7 defined as normal case, scored 8 to 10 defined as doubtful case, and scored 11 to 21 defined as definite case. The proportion of definite anxiety cases of the two study arms will be compared.
Proportion of definite depression cases | This outcome will be assessed right before the next scheduled clinic for histological results (around 1 to 2 weeks after polypectomy)..
  The level of depression of the two study arms will be measured by using the Taiwan version questionnaire of Hospital Anxiety and Depression Scale (HADS) right before the next scheduled clinic for histological results. The depression score of this questionnaire ranging from 0 to 21. Scored 0 to 7 defined as normal case, scored 8 to 10 defined as doubtful case, and scored 11 to 21 defined as definite case. The proportion of definite depression cases of the two study arms will be compared.

SECONDARY OUTCOMES:
Anxiety score | This outcome will be assessed right before the next scheduled clinic for histological results (around 1 to 2 weeks after polypectomy)..
  The level of anxiety of the two study arms will be measured by using the Taiwan version questionnaire of Hospital Anxiety and Depression Scale (HADS) right before the next scheduled clinic for histological results and compared the difference between the two study arms. The anxiety score of this questionnaire ranging from 0 to 21. Higher score means higher anxiety level.
Depression score | This outcome will be assessed right before the next scheduled clinic for histological results (around 1 to 2 weeks after polypectomy)..
  The level of depression of the two study arms will be measured by using the Taiwan version questionnaire of Hospital Anxiety and Depression Scale (HADS) right before the next scheduled clinic for histological results and compared the difference between the two study arms. The depression score of this questionnaire ranging from 0 to 21. Higher score means higher depression level.

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giorgi Rossi P, Vicentini M, Sacchettini C, Di Felice E, Caroli S, Ferrari F, Mangone L, Pezzarossi A, Roncaglia F, Campari C, Sassatelli R, Sacchero R, Sereni G, Paterlini L, Zappa M. Impact of Screening Program on Incidence of Colorectal Cancer: A Cohort Study in Italy. Am J Gastroenterol. 2015 Sep;110(9):1359-66. doi: 10.1038/ajg.2015.240. Epub 2015 Aug 25. PMID 26303133
- [Background] Chiu HM, Chen SL, Yen AM, Chiu SY, Fann JC, Lee YC, Pan SL, Wu MS, Liao CS, Chen HH, Koong SL, Chiou ST. Effectiveness of fecal immunochemical testing in reducing colorectal cancer mortality from the One Million Taiwanese Screening Program. Cancer. 2015 Sep 15;121(18):3221-9. doi: 10.1002/cncr.29462. Epub 2015 May 20. PMID 25995082
- [Background] Denters MJ, Deutekom M, Bossuyt PM, Fockens P, Dekker E. Patient burden of colonoscopy after positive fecal immunochemical testing for colorectal cancer screening. Endoscopy. 2013;45(5):342-9. doi: 10.1055/s-0032-1326238. Epub 2013 Mar 12. PMID 23483433
- [Background] Denters MJ, Deutekom M, Essink-Bot ML, Bossuyt PM, Fockens P, Dekker E. FIT false-positives in colorectal cancer screening experience psychological distress up to 6 weeks after colonoscopy. Support Care Cancer. 2013 Oct;21(10):2809-15. doi: 10.1007/s00520-013-1867-7. Epub 2013 Jun 1. PMID 23729229
- [Background] Oba S, Tanaka S, Sano Y, Oka S, Chayama K. Current status of narrow-band imaging magnifying colonoscopy for colorectal neoplasia in Japan. Digestion. 2011;83(3):167-72. doi: 10.1159/000321807. Epub 2011 Jan 21. PMID 21266811
- [Background] Sumimoto K, Tanaka S, Shigita K, Hayashi N, Hirano D, Tamaru Y, Ninomiya Y, Oka S, Arihiro K, Shimamoto F, Yoshihara M, Chayama K. Diagnostic performance of Japan NBI Expert Team classification for differentiation among noninvasive, superficially invasive, and deeply invasive colorectal neoplasia. Gastrointest Endosc. 2017 Oct;86(4):700-709. doi: 10.1016/j.gie.2017.02.018. Epub 2017 Feb 28. PMID 28257790
- [Background] Matsuda T, Fujii T, Saito Y, Nakajima T, Uraoka T, Kobayashi N, Ikehara H, Ikematsu H, Fu KI, Emura F, Ono A, Sano Y, Shimoda T, Fujimori T. Efficacy of the invasive/non-invasive pattern by magnifying chromoendoscopy to estimate the depth of invasion of early colorectal neoplasms. Am J Gastroenterol. 2008 Nov;103(11):2700-6. doi: 10.1111/j.1572-0241.2008.02190.x. Epub 2008 Oct 3. PMID 18853968
- [Background] Mason SE, Poynter L, Takats Z, Darzi A, Kinross JM. Optical Technologies for Endoscopic Real-Time Histologic Assessment of Colorectal Polyps: A Meta-Analysis. Am J Gastroenterol. 2019 Aug;114(8):1219-1230. doi: 10.14309/ajg.0000000000000156. PMID 30848728
- [Background] Backes Y, Moss A, Reitsma JB, Siersema PD, Moons LM. Narrow Band Imaging, Magnifying Chromoendoscopy, and Gross Morphological Features for the Optical Diagnosis of T1 Colorectal Cancer and Deep Submucosal Invasion: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2017 Jan;112(1):54-64. doi: 10.1038/ajg.2016.403. Epub 2016 Sep 20. PMID 27644737
- [Background] ASGE Technology Committee; Abu Dayyeh BK, Thosani N, Konda V, Wallace MB, Rex DK, Chauhan SS, Hwang JH, Komanduri S, Manfredi M, Maple JT, Murad FM, Siddiqui UD, Banerjee S. ASGE Technology Committee systematic review and meta-analysis assessing the ASGE PIVI thresholds for adopting real-time endoscopic assessment of the histology of diminutive colorectal polyps. Gastrointest Endosc. 2015 Mar;81(3):502.e1-502.e16. doi: 10.1016/j.gie.2014.12.022. Epub 2015 Jan 16. PMID 25597420
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820